CLINICAL TRIAL: NCT00005918
Title: The Safety and Antiviral Efficacy of Stavudine Extended Release Formulation as Compared to Stavudine Immediate Release Formulation, Each as Part of Potent Antiretroviral Combination Therapy
Brief Title: Effectiveness and Safety of Two Forms of Stavudine in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 244F; AI455-099
Record Dates: First submitted 2000-06-15; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Stavudine; Lamivudine; RNA, Viral; Dosage Forms; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Efavirenz
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of 2 forms of stavudine (d4T). One form is taken once a day (extended release) and the other form is taken twice a day (immediate release).

DETAILED DESCRIPTION:
Patients are randomized to receive blinded stavudine extended release (d4T ER) or immediate release (d4T IR) formulation. Randomization is balanced by screening HIV viral load of less than 30,000 copies/ml or at least 30,000 copies/ml and by site. Patients also receive open-label efavirenz (EFV) and lamivudine (3TC). Efficacy is evaluated over 48 weeks of the dosing period and safety is evaluated over the entire dosing period (56 weeks).

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old. Patients living in USA, Puerto Rico, Australia, Brazil, Singapore, and Thailand can be at least 12 years old (need consent of parent or guardian if under 18).
* Have a viral load of at least 2,000 copies/ml within 21 days of study entry.
* Have a CD4 count of at least 100 cells/mm3 within 21 days of study entry.
* Agree to use a barrier method of birth control (such as condoms) during the study.
* Are available for follow-up for at least 56 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have taken nonnucleoside reverse transcriptase inhibitors (NNRTIs) or protease inhibitors (PIs) for more than 30 days and within 14 days of study entry.
* Have a new opportunistic (HIV-related) infection or condition requiring treatment.
* Have acute (early) HIV infection.
* Have diarrhea (at least 6 loose stools/day for at least 7 days in a row) within 30 days prior to study entry.
* Abuse alcohol or drugs.
* Have active hepatitis within 30 days prior to study entry.
* Have a history of peripheral neuropathy (a condition affecting the nervous system).
* Cannot take medications by mouth.
* Are allergic to certain antiviral drugs.
* Need to take certain medications that should not be taken with EFV.
* Have certain other conditions or prior treatments that might affect the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 730
Dates: Start 2000-06; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (18):
  - AIDS Healthcare Foundation, Los Angeles, California
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Med Alternatives, Fort Lauderdale, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - The CORE Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Univ of Louisville, Louisville, Kentucky
  - CRI of New England, Brookline, Massachusetts
  - CRI - Springfield, Springfield, Massachusetts
  - No Nevada HOPES, Reno, Nevada
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ Hospital, Oklahoma City, Oklahoma
  - Aesculapisu Medical Health Group, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Plaza Med Ctr, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
- Argentina (8):
  - Arnaldo Casiro MD, Buenos Aires
  - Claudia Rodriguez MD, Buenos Aires
  - Elida Pallone MD, Buenos Aires
  - Fundacion Huesped, Buenos Aires
  - Luis Maria Zieher MD, Buenos Aires
  - Fernando Silva Nieto MD, Prov Bs As
  - CAICI, Rosario Santa Fe
  - Marcelo Beltran, San Isidro
- Australia (2):
  - Hugo Ree MD, Brisbane
  - Prahran Market Clinic, South Yarra
- Belgium (2):
  - University Hospital Gent, Ghent
  - Domaine Universitaire Du SART-TILMAN, Liège
- Brazil (5):
  - Federal University of Minas, Dept. of Pediatrics, Belo Horizonte-MG
  - Universidade Estadual de Botucatu, Botucatu-SP
  - Ricardo Leite Hayden, Santos
  - Fundacao Zerbini Casa Da Aids, São Paulo
  - Instituto de Infectologia Emilio Ribas, São Paulo
- Canada (4):
  - Saint Paul's Hosp, Vancouver, British Columbia
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Dr Roger P Leblanc, Montreal, Quebec
- France (5):
  - Hopital Saint Andre, Bordeaux
  - Hopital Edouard Herriot, Lyon
  - Hopital De L'Hotel Dieu, Nantes
  - Srev Du Pr Gentilini, Paris
  - Hopital Pontachaillou, Rennes
- Israel (2):
  - Kaplan Med Ctr, Rehovot
  - Sheba Med Ctr, Tel Litwinsky
- Italy (8):
  - Reparto Malattie Infettive, Antella
  - Universita Di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - Ospedale Luigi Cacco Moroni, Milan
  - Ospedale Cotugno, Napoli
  - Ospedale Cisanello, Pisa
  - Ospedale Amedeo de Savoia, Torino
  - Ospedale Amedeo di Savoia, Torino
- Mexico (4):
  - Hospital General, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City
  - Instituto Nacional de la Nutricion, Mexico City
  - Alberto Orneals MD, Tijuana
- Portugal (3):
  - Hospital Distrital de Almada, Almada
  - Hospital Universidade De Coimbra, Coimbra
  - Hosp De Santa Maria, Lisbon
- Puerto Rico (2):
  - San Cristobal Hosp, Coto Laurel, Ponce
  - Clinical Research Puerto Rico Inc, San Juan
- Russia (2):
  - Federal AIDS Ctr, Moscow
  - Nina Volkova MD, Saint Petersburg
- South Africa (5):
  - Tygerberg Hosp, Cape Town
  - Chris Hani Baragwanath Hosp, Johannesburg
  - Innovir Institute / Saffer House, Johannesburg
  - Johannesburg Hosp, Johannesburg
  - Embassy Drive Medical Centre, Pretoria
- Spain (4):
  - Hosp Clinic, Barcelona
  - Hosp Gregorio Maranon, Madrid
  - Hosp son Dureta, Palma de Mallorca
  - Hosp de Navarra, Pamplona
- Thailand (2):
  - Chulalongkorn Univ Hosp / HIV / NAT Rsch Collab, Bangkok
  - Bamrasnaradura Hosp, Nontaburi
- Tan tock Seng Hosp